CLINICAL TRIAL: NCT04880408
Title: Morphological and Metabolic Changes of Dorsal Root Ganglion and Sympathetic Ganglion in Patients With Postherpetic Neuralgia on MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianwei Zhang，MD, Clinical Professor, Huazhong University of Science and Technology
Other Study IDs: herpes zoster
Record Dates: First submitted 2021-04-22; First posted 2021-05-10 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Pain; Neuropathy;Peripheral
Keywords: herpes zoster; postherpetic neuralgia; MRI; dorsal root ganglion
MeSH Terms: conditions — Pain; Neuritis; Herpes Zoster; Neuralgia, Postherpetic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Object: Postherpetic neuralgia (PHN) is pain that persists for 1-3 months after herpes zoster onset. It is the most common complication of herpes zoster and occurs in 15-40% of patients with herpes zoster. PHN has been suggested to be related with the lesion of doral root ganglion (DRG). However, the studies are almost limited to autopsies and animals , and the mechanism of PHN is still unclear. This study was conducted to investigate morphological and metabolic changes of DRG and sympathetic ganglion in patients with postherpetic neuralgia on MRI. Method: 30 patients diagnosed as PHN were recruited. The volume and fractional anisotropy of DRG of lesion dermatomes were measured under MRI, and compared with contralateral and adjacent DRG. The volume and fractional anisotropy of sympathetic ganglion of lesion dermatomes were also measured under MRI, and compared with contralateral and adjacent sympathetic ganglion.Then, the association between clinical phenotypes and DRG changes were analyzed.

DETAILED DESCRIPTION:
Patients with the following conditions were excluded: psychiatric diseases or communication disorders; contraindications to MRI;DRG radiofrequency therapy, spinal cord electrical stimulation and other direct intervention treatments for DRG were performed before examination.

ELIGIBILITY:
Inclusion Criteria:

* aged more than 18 herpes zoster in cervical, thoracic,lumbar or sacral regions agree to participate to the research

Exclusion Criteria:

* can not cooperate to MRI for mental disease contraindication for MRI treatments for DRG such as radiaofrequency therapy, spinal cord electircal stimulation were performed before examination. disagree to participate to the research

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with herpes zoster in cervical, thoracic,lumbar or sacral regions
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
To compare the volume and fractional anisotropy of DRG between lesion dermatomes and contralateral dermatomes | 1 year
  DRGs of lesion and contralateral dermatomes were scanned under MRI. Then, the valume (the maximum cross-section area ×layers/2) and fractional anisotropy of DRGs were measured with RadiAnt DICOM Viewer, and the comparison was made between lesion and contralateral DRG.

SECONDARY OUTCOMES:
To compare the volume and fractional anisotropy of sympathetic ganglion between lesion dermatomes and contralateral dermatomes. | 1 year
  as primary outcome measure, sympathetic ganglions of lesion and contralateral dermatomes were scanned under MRI. Then, the valume (the maximum cross-section area ×layers/2) and fractional anisotropy of sympathetic ganglions were measured with RadiAnt DICOM Viewer, and the comparison was made between lesion and contralateral sympathetic ganglions.
To compare the volume and fractional anisotropy of DRG between lesion dermatomes and adjacent dermatomes. | 1 year
  DRGs of lesion and adjacent dermatomes were scanned under MRI. Then, the valume (the maximum cross-section area ×layers/2) and fractional anisotropy of DRGs were measured with RadiAnt DICOM Viewer, and the comparison was made between lesion and adjacent DRG.

CONTACTS AND LOCATIONS:
Overall Officials: Xianwei Zhang, Doctor, Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China